CLINICAL TRIAL: NCT01438671
Title: Does Wii Fit Balance Training Significantly Improve Standing Balance Compared to Traditional Balance Training and Is Wii Fit Balance Training Preferred Over Traditional Balance Training by Patients With SCI/TBI/CVA?
Brief Title: Wii Fit Balance Training Compared to Traditional Balance Training in Patients With SCI/TBI/CVA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Facility where study was taking place closed.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1179437
Record Dates: First submitted 2011-08-02; First posted 2011-09-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Distorted; Balance
Keywords: WiiFit; Standing Balance; Neurological Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): Nintendo Wii Fit Balance training followed by traditional balance training
  Interventions: Procedure: Nintendo Wii Fit; Procedure: Traditional balance training

INTERVENTIONS:
Procedure: Nintendo Wii Fit — The Nintendo Wii Fit is an accessory for the Nintendo Wii video game system that utilizes a balance board peripheral. The subject stands on the balance board and engages in video games that require weight shifting and balancing in order to interact with the game. This intervention will be administered for 30 minutes, 3 to 5 times per week (as tolerated by subject), for a two week period.
Procedure: Traditional balance training — This physical therapy intervention involves gait training, balance education on various surfaces, activities involving limited and changing bases of support, and dynamic interaction with the subject's environment. This intervention will be administered 30 minutes per day, 3 to 5 days per week (by subject's tolerance), for a two week period.

SUMMARY:
Our hypothesis is the investigators will find a significant advantage for the use of a virtual reality system like the Wii Fit to improve overall balance scores versus the use of traditional balance activities alone. The objectives will be to determine the enjoyment of these types of gaming activities through the use of a survey to support the hypothesis that these activities are more enjoyable than traditional activities and to gather evidence to support the use of these more enjoyable activities as a viable and needed addition to the overall balance regimen given in the plan of care for a patient with traumatic or acquired brain injury, stroke or spinal cord injury.

DETAILED DESCRIPTION:
In the recent past and currently, the Wii Fit has been and will probably continue to be used as an effective rehabilitation aide in improving balance and coordination in all populations. It is another tool amongst traditional balance activities to assist the therapist and patient in reaching the goals of both parties and improving overall functional outcomes for the patient. The Wii Fit is capable of giving objective data in a stimulating environment in which to deliver fun yet effective and measurable balance training. The addition of fun and enjoyment is found in most populations using a virtual reality system like the Wii. (VR Rehab, 2008) Brumels et al suggested having lack of interest in an activity can lead to less than desired engagement and performance (Comparison, 2008), which can lead to overall less improvement. This was supported at the conclusion of their study, indicating scientific reason to include the use of video game based programs in clinical settings. If someone is interested in a task because it is enjoyable and it keeps their interest over and over then, because of the increased time practicing due to the desire to actually participate, they are more inclined to make improvements in the task being practiced. In the case of this study, balance would be the task improving.

However, the same investigators concluded further research is required in order to determine the utility of an off-the-shelf gaming system like the Wii. One purpose of this project is to determine the effectiveness of this type of system with the hopes of eventually working with a company like Nintendo to make adjustments to their software and hardware systems in order to provide a comprehensive and adaptive system to deliver balance re-education to multiple populations. We also would like to determine, through the use of participant satisfaction surveys, if individuals prefer the use of a system like the Wii Fit over traditional balance exercises since improvements in balance can be linked to improved participation based on the enjoyment of the activity. If we can show that both the Wii Fit system itself is a viable apparatus with which to address and improve balance outside of traditional balance activities and that participants enjoy this method of balance activities then we open up the opportunity for a larger number of ways to assist in balance recovery for those affected with some sort of balance deficit. As the study by S M Flynn, et al, concluded, the use of systems like the WiiFit may encourage individuals to "play" with and against others promoting a healthier and less isolating lifestyle.

The clinical trials in this study will be conducted in compliance with the mentioned protocol and within the regulations set by the University of Missouri and the Missouri Rehabilitation Center. The population to be studied will be individuals from the ages of 16-70 with varying degrees of functional abilities after traumatic or acquired brain injury, stroke or spinal cord injury who do possess the physical capabilities as explained in the below inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Acquired neurological diagnosis
* 18 years of age or greater
* Score greater than or equal to an 18 on the MME and/or have a FIM score of 5 in comprehension and problem solving.
* Ability to stand with no greater than minimal assist (FIM score of 4, less than or equal to 25% assist)
* Vision that is WFL with or without glasses/contacts
* Ability to stand for at least 5 minutes without rest.
* Have at least a WBAT status

Exclusion Criteria:

* Person that is less than 18 years of age
* Person scoring less than an 18 on the MME and/or a FIM score of a 4 or lower in comprehension and problem solving.
* Person with the inability to stand without minimal assist
* Inability to stand for 5 minutes without rest
* Impaired vision
* Weight bearing precautions of 50%WB or NWB on either lower extremity
* Any vestibular diagnoses
* Pain that limits participation
* Uncontrollable medical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
WiiFit | Before and after two consecutive 2 week periods: one period without intervention, one with
  For standing balance we will be using the Berg Balance Scale and Single Leg Stance.
  The investigators will also be looking at weight bearing symmetry utilizing the intrinsic tests included with the Nintendo Wii Fit ™ Measurements will be taken at baseline (pre-intervention), and at conclusion of each intervention phase (after 2 weeks of traditional balance therapy and then again after 2 weeks of training using the Nintendo Wii Fit ™)

SECONDARY OUTCOMES:
Satisfaction | Post Intervention (at conclusion of two 2 week trials)
  For patient preferences in intervention we will be using the Intrinsic Motivation Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey D. Mosley, PT, Principal Investigator — Missouri Rehabilitation Center, University of Missouri Health Systems
Locations (1):
- Missouri Rehabilitation Center, Mount Vernon, Missouri, United States

IPD SHARING:
Plan to Share IPD: No